CLINICAL TRIAL: NCT04013516
Title: Measles Vaccination Cash Incentives Experimental Evidence From Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDinsight (Other)
Collaborators: GiveWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 004
Record Dates: First submitted 2019-06-27; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Measles
Keywords: Immunization; Incentives
MeSH Terms: conditions — Measles | interventions — CD56 Antigen

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to different incentive amounts (treatment arms), a pure control arm, and a placebo arm which consisted of a phone call without an additional incentive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pure Control (No Intervention): Respondents received New Incentives' normal program.
- Reminder Call (Placebo Comparator): Respondents received a call from a New Incentives' staff member similar to the treatment arms, but weren't offered additional incentives.
  Interventions: Behavioral: Call
- Small Additional Incentive (Experimental): Respondents were told they would receive 1000 NGN more than originally promised by New Incentives' (either 2000 or 3000 NGN) when they brought their child for measles immunization.
  Interventions: Behavioral: Cash Incentive; Behavioral: Call
- Large Additional Incentive (Experimental): Respondents were told they would receive 3000 NGN more than originally promised by New Incentives' (either 2000 or 3000 NGN) when they brought their child for measles immunization.
  Interventions: Behavioral: Cash Incentive; Behavioral: Call

INTERVENTIONS:
Behavioral: Cash Incentive — During the phone call, New Incentives' team member promised a greater cash payment from New Incentives' staff members at primary health care facilities when infants enrolled in the program and received their measles vaccination.
  Arms: Large Additional Incentive; Small Additional Incentive
Behavioral: Call — A New Incentives' team member reminded caregivers of their child's measles immunization date and the total amount of incentive they would receive once their child was vaccinated. If the caregiver could not be reached on the first attempt, the team made additional attempts at different times of the day on five different days across two weeks (up to 10 attempts were made per caregiver).
  Arms: Large Additional Incentive; Reminder Call; Small Additional Incentive

SUMMARY:
IDinsight is conducting a randomized controlled trial to assess the impact of various sized cash incentives for caretakers of infants that require a 9-month measles vaccination on the completion rate for the vaccine in Nigeria. The purpose of the experiment is to help New Incentives (NI) determine the optimal size of the incentive as they scale to the North West region of Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver and infant registered with the New Incentives program
* The infant was nine months or older at the start of the study (note there was no upper age limit as New Incentives only began enrolling infants in October 2016)
* Infant had received at least one previous conditional cash transfer for immunization at an All Babies are Equal Initiative clinic,
* Infant had received their Penta-3 vaccine.
* The caregiver had provided a phone number (either a personal number or a number of someone who can reach them) during registration.

Exclusion Criteria:

* Infant had already received a measles vaccine

Min Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1088 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Measles Vaccination Coverage Rate | We assessed whether eligible infants received measles vaccination at any time during the 4 month study period. Children were a minimum of 9 months at the beginning of the study and a maximum of 7 years at the end of the study.
  The outcome of interest is the measles coverage rate among the eligible randomized infants. Coverage is measured using the measles vaccination information recorded on the child's health card. The child health card information was immediately entered into the New Incentives' database by their field staff when they disbursed the cash incentives at program clinics. Information from the New Incentives' database was used for the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Connor, Principal Investigator — IDinsight
Locations (1):
- All Babies are Equal Initiative (New Incentives), Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Include anonymized data and study protocol as supplementary materials for the published article.
Supporting Information: Study Protocol
Time Frame: At the time of publication.